CLINICAL TRIAL: NCT00483483
Title: Maximizing Opportunity: HIV Prevention in Hospitalized Russian Drinkers
Brief Title: Project HERMITAGE: HIV Prevention in Hospitalized Russian Drinkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Jeffrey Samet, Chief, Section of General Internal Medicine, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-25082; R01AA016059 (NIH)
Record Dates: First submitted 2007-06-06; First posted 2007-06-07 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: HIV Infections
Keywords: HIV; Unsafe sex; High-risk sex; Needle sharing; STDs
MeSH Terms: conditions — HIV Infections; Unsafe Sex; Sexually Transmitted Diseases | interventions — Self-Help Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): Healthy Relationships Intervention (HRI)
  Interventions: Behavioral: Individual and group HIV risk behavior counseling sessions
- Attention-control group (Active Comparator): health education & support
  Interventions: Behavioral: health education and support group

INTERVENTIONS:
Behavioral: Individual and group HIV risk behavior counseling sessions — Healthy Relationships Intervention (HRI) culturally adapted and modified to address substance use and associated risk behaviors; subjects will attend three 2-hour structured group sessions in addition to two 1-hour individualized sessions over the course of 10 days.
  Other Names: HRI
  Arms: 1
Behavioral: health education and support group — general health information (nutrition, stress reduction) in 2 individual sessions and 3 group sessions.
  Arms: Attention-control group

SUMMARY:
The objective of this study is to test in a randomized controlled trial the effectiveness of a US secondary HIV prevention program to reduce HIV risk behaviors, STD acquisition, and alcohol consumption among HIV-infected Russians with risky drinking.

DETAILED DESCRIPTION:
Russia has one of the fastest growing AIDS epidemics in the world, with an estimated 1 million HIV-infected persons. Initially the Russian HIV epidemic was almost exclusively among injection drug users (IDUs); however, concern exists that HIV is expanding into the general population via sexual transmission. Alcohol use, highly prevalent in Russia, may increase high-risk sexual behaviors among IDUs and alcohol dependent persons. Furthermore, animal models suggest that alcohol consumption plays a permissive role for HIV replication as the resultant higher viral loads may increase risk of transmission. Thus alcohol use may accelerate HIV transmission to the general population in Russia.

The study will randomize 700 HIV-infected patients with risky alcohol consumption to an adapted Healthy Relationships Intervention (HRI) or attention-control support groups. The intervention will be culturally adapted and modified to address substance use and associated risk behaviors. Subjects participating in the HRI will attend three 90-120 min structured group sessions in addition to two 30-60 min individualized sessions over the course of 5-10 days. Subjects in the attention-control group will participate in general health information sessions in the same format (i.e., 2 individualized and 3 group sessions) during the same timeframe.

All patients will be assessed at baseline (pre-randomization) and 6-months and 12-months post-randomization at the recruitment site. Primary outcomes are HIV sex and drug risk behaviors and sexually transmitted diseases. Additionally, subjects will be assessed regarding secondary outcomes including alcohol consumption, quality of life and social support, victimization, suicide, overdose, and disclosure of HIV serostatus.

We hypothesize that relative to the comparison group, participants receiving the adapted Healthy Relationships Intervention will have reduced HIV sex and drug risk behaviors and STD acquisition. If the intervention is effective among HIV-infected hospitalized patients, it could be used to address other HIV infected persons in a variety of Russian settings potentially reducing the transmission of HIV by decreasing risky sex and drug use behaviors among Russians.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years old;
* HIV positive;
* Alcohol consumption at NIAAA at-risk drinking levels (greater than 14 drinks per week [or more than 4 drinks per day] for men, and greater than 7 drinks per week [or more than 3 drinks per day] for women) during the 30 days prior to hospital admission, For subjects whose drinking was not risky 30 days prior to hospital admission, we will ask if their drinking was equivalent to binge amounts on any day in the prior 6 months;
* Self-reported unprotected anal or vaginal sex in the last 6 months;
* Provision of contact information (e.g., name, home address, telephone number) of two relatives or close friends who can be contacted to share information that may be used to assist with follow-up;
* Stable address within St. Petersburg or districts within 150 kilometers of St. Petersburg; and
* Possession of a home telephone;
* Fluent in Russian;
* Ability to provide informed consent.

Exclusion Criteria:

* Severe cognitive impairment (i.e., clinically apparent dementia, active psychosis, or severe paranoid disorder) as judged by a hospital clinician and stated in the records;
* Acute illness precluding ability to participate in assessment for eligibility (however these patients may be assessed again on a subsequent day);
* Trying to get (partner) pregnant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2007-10; Primary Completion 2011-07 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Number of unprotected sex acts, unclean drug injections, and sexually transmitted infections (by urinalysis) | 12 months

SECONDARY OUTCOMES:
Percentage of protected sex episodes, percentage of unprotected sex episodes Multiple drug partners, Number of sexually transmitted infections (by self report), Alcohol consumption, Disclosure of HIV serostatus | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey H. Samet, MD, MA, MPH, Principal Investigator — Boston Medical Center, Boston University
Locations (3):
- Russia (3):
  - City Drug Addiction Center, Saint Petersburg
  - Pavlov State Medical University and Botkin Infectious Disease Hospital, Saint Petersburg
  - St. Petersburg AIDS Center, Saint Petersburg

REFERENCES:
- [Derived] Greene MC, Kane J, Alto M, Giusto A, Lovero K, Stockton M, McClendon J, Nicholson T, Wainberg ML, Johnson RM, Tol WA. Psychosocial and pharmacologic interventions to reduce harmful alcohol use in low- and middle-income countries. Cochrane Database Syst Rev. 2023 May 9;5(5):CD013350. doi: 10.1002/14651858.CD013350.pub2. PMID 37158538
- [Derived] Samet JH, Blokhina E, Cheng DM, Walley AY, Lioznov D, Gnatienko N, Quinn EK, Bridden C, Chaisson CE, Toussova O, Gifford AL, Raj A, Krupitsky E. A strengths-based case management intervention to link HIV-positive people who inject drugs in Russia to HIV care. AIDS. 2019 Jul 15;33(9):1467-1476. doi: 10.1097/QAD.0000000000002230. PMID 30964750
- [Derived] Lunze K, Lioznov D, Cheng DM, Nikitin RV, Coleman SM, Bridden C, Blokhina E, Krupitsky E, Samet JH. HIV Stigma and Unhealthy Alcohol Use Among People Living with HIV in Russia. AIDS Behav. 2017 Sep;21(9):2609-2617. doi: 10.1007/s10461-017-1820-8. PMID 28600603
- [Derived] Samet JH, Raj A, Cheng DM, Blokhina E, Bridden C, Chaisson CE, Walley AY, Palfai TP, Quinn EK, Zvartau E, Lioznov D, Krupitsky E. HERMITAGE--a randomized controlled trial to reduce sexually transmitted infections and HIV risk behaviors among HIV-infected Russian drinkers. Addiction. 2015 Jan;110(1):80-90. doi: 10.1111/add.12716. Epub 2014 Oct 16. PMID 25170994